CLINICAL TRIAL: NCT05140291
Title: Dry Needling of the Trigeminal Nerve Innervation Field for Cervicogenic Eadache: A Pilot Study
Brief Title: Dry Needling for Cervicogenic Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Youngstown State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-6
Record Dates: First submitted 2021-10-29; First posted 2021-12-01 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Double blinded, sham controlled, randomized trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be asked to keep their eyes closed during the treatment. Clinicians will be blinded to group and outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Experimental Group
  Interventions: Other: Dry Needling
- Sham Needling (Sham Comparator): Sham Group
  Interventions: Other: Sham Dry Needling

INTERVENTIONS:
Other: Dry Needling — 1/2" needles will placed into defined innervation fields of the trigeminal nerve and rotated. Total time will be 5-7 minutes.
  Arms: Dry needling
Other: Sham Dry Needling — Needle handles inside of guide tubes will be tapped in a way similar to an actual needle being set but the sham needles will be blunted.
  Arms: Sham Needling

SUMMARY:
Currently, it is unknown if dry needling when performed to the trigeminal innervation field improves neck pain and or headache for patients with cervicogenic headaches. The aim of this study is to determine if dry needling of the trigeminal innervation field improves pain, pain-pressure thresholds, and neck mobility in patients with cervicogenic headaches, with or without migraine.

DETAILED DESCRIPTION:
Dry needling is a widely used intervention performed by physical therapists for a wide range of musculoskeletal and neurological conditions. Dry needling has been shown to be beneficial for cervicogenic headaches but treatment is typically applied to the neck. It is well-established that cervical pain can upregulate the trigeminal nerve and vice versa in various forms of headaches. Thus, it is plausable that reducing inflammation and irritation of the trigeminal nerve may in fact reduce neck pain and impairments. This study aims to look investigate whether dry needling the trigeminal innervation field will reduce pain and impairments known to exist in patients with cervicogenic headaches compared to a sham comparator. The study is a pilot trial for a larger RCT and will look at immediate effects only.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Symptoms: (1)Unilateral pain starting in the neck and radiating to the frontotemporal region or posterior fossa, (2) pain aggravated by neck movement, (3) restricted cervical range of motion, (4) non-throbbing and non-lancinatingnpain, 5) dysfunction/headache pain in at least one of the joints of the upper cervical spine(C0-C4), and (6) headache frequency of at least 1 per week over a period greater than 3 months.

Exclusion Criteria

* Pain <2/10
* Contraindications to the interventions
* Whiplash associated disorder within 6 weeks
* Pending litigation for neck pain and/or headache.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Headache or neck pain intensity on a Numeric pain rating scale (0-10) | <1 hour
  0-10 scale pain intensity

SECONDARY OUTCOMES:
Active Range of Motion of the Cervical Spine in degrees of measurement | <1 hour
  Active range of motion will be measured in the most painful and or limited plane of movement.
Flexion-rotation test in degrees of measurement | <1 hour
  Flexion-rotation test for CGH will be measured to determine any change in measure for c1-c2 mobility.
Pain-pressure threshold in lbs of pressure | <1 hour
  Pain-pressure threshold will be measured using an algometer at the innervation zones of the trigeminal nerve and the upper cervical spine.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Lieber, PhD, Study Director — Director of the PhD in Health Sciences
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vazquez-Justes D, Yarzabal-Rodriguez R, Domenech-Garcia V, Herrero P, Bellosta-Lopez P. Effectiveness of dry needling for headache: A systematic review. Neurologia (Engl Ed). 2020 Jan 13:S0213-4853(19)30144-6. doi: 10.1016/j.nrl.2019.09.010. Online ahead of print. English, Spanish. PMID 31948718
- [Background] Gildir S, Tuzun EH, Eroglu G, Eker L. A randomized trial of trigger point dry needling versus sham needling for chronic tension-type headache. Medicine (Baltimore). 2019 Feb;98(8):e14520. doi: 10.1097/MD.0000000000014520. PMID 30813155
- [Background] France S, Bown J, Nowosilskyj M, Mott M, Rand S, Walters J. Evidence for the use of dry needling and physiotherapy in the management of cervicogenic or tension-type headache: a systematic review. Cephalalgia. 2014 Oct;34(12):994-1003. doi: 10.1177/0333102414523847. Epub 2014 Mar 12. PMID 24623124